CLINICAL TRIAL: NCT06654427
Title: Trauma-Informed Obstetric Care: Development and Implementation of a Stakeholder- Informed Toolkit for Obstetric Providers and Patients
Brief Title: Trauma-Informed Obstetric Care: Development and Implementation of a Toolkit for Obstetrics (OBTIC)
Acronym: OBTIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: K23HD107296-01A1 (NIH)
Record Dates: First submitted 2023-07-09; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Trauma; Obstetrics Trauma; Pregnancy Related
Keywords: trauma informed care; Obstetrics
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The OBTIC toolkit will be used in an obstetrics clinic for a 9 month period. Baseline will be evaluated 3 months pre-implementation trial and follow-up will be measured 3 months post-implementation trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of OBTIC (Experimental): The OB-TIC intervention toolkit will be pilot tested in outpatient obstetrics clinics. OB-TIC will be implemented for 9 months during which time I will assess providers' and patients' perceptions of acceptability, appropriateness, and feasibility of OB-TIC. Adoption of OB-TIC, attitudes towards TIC, appointment adherence and care choices, maternal-infant health outcomes, and patient mental health will be assessed before, during, and after the pilot.
  Interventions: Behavioral: Obstetric Trauma Informed Care Toolkit

INTERVENTIONS:
Behavioral: Obstetric Trauma Informed Care Toolkit — The OB-TIC toolkit will include provider and staff training on trauma- informed care and information on trauma-related perinatal concerns; trauma assessment tools; trauma-informed procedure modifications; clinical language guides; patient-facing resources including birth strategies, referral resources, and education; and clinical language. The OB-TIC intervention will utilize the toolkit to integrate trauma-informed care into clinical practice. Implementation strategies will be assessed to determine the most effective method for integrating OB-TIC content into practice.
  Other Names: OBTIC; STAR-OB

SUMMARY:
Many pregnant women have experienced trauma, which can make perinatal care stressful and increase the risk of pregnancy-related health conditions. However, obstetric providers can modify procedures to reduce distress and enhance patients' sense of control and safety. Although obstetric providers frequently care for trauma survivors, most are not trained in trauma-informed care (TIC). Additionally, there are no data on feasibility, appropriateness, or acceptability of TIC tools and interventions in the context of obstetrics. The goal of this project is to develop the first, stakeholder-informed obstetric TIC toolkit composed of treatment protocols, clinician training, trauma and violence screening tools, and other resources to help obstetric providers apply TIC practices to all clinical interactions in addition to identifying and providing support for trauma survivors. The obstetric TIC intervention toolkit (OB-TIC) will be developed in collaboration with key stakeholders (pregnant and postpartum patients, nurses, physicians, and administrators) to ensure that it is feasible, acceptable, appropriate, cost-effective, and clinically useful. Current practices and preferences will be characterized in qualitative interviews with stakeholders which will inform the development of OB-TIC in collaboration with a community working group of stakeholders. A pilot implementation trial of OB-TIC will be conducted in two outpatient obstetrics clinics to gather real-world data that will inform the final intervention toolkit, which will be tested on a larger scale in future studies.

DETAILED DESCRIPTION:
The goal of this study is to develop a stakeholder-informed toolkit for obstetric providers and patients to support the implementation of trauma-informed care (TIC) in routine clinical practice. Following interviews with providers and pregnant/postpartum participants as well as convening with a community working group of stakeholders, an OBTIC toolkit blueprint will be drafted for testing.

In the pilot implementation phase, all clinicians and administrators at an outpatient obstetrics clinic will participate in the OB-TIC intervention. However, only providers who consent to participate in surveys and interviews will be contacted by the PI to complete surveys (assessment of attitudes related to TIC and usefulness of toolkit components) at the mid-point (month 2) and after completion of the pilot (month 4). Clinicians will also be interviewed as a group (physicians and nurses separately) following a staff meeting; interviews will assess perceived acceptability, feasibility, appropriateness and helpfulness of the toolkit. Additionally, 12-20 postpartum participants, who were treated at the clinic during the pilot, will be recruited for brief semi-structured qualitative interviews and surveys following the completion of the pilot (see detail in 2.5). In order to assess adoption of the trauma screening component of the TIC toolkit, I will conduct chart review of initial prenatal visits at baseline (3 months prior) during (9 months of the pilot trial) and after completion (3 months following completion) of the pilot trial to assess rates of screening. To assess exploratory efficacy outcomes, I will use chart review to collect data on 1) Perinatal care: care engagement (appointment adherence, attendance of postpartum follow-up), and care choices (elective augmentation of delivery); 2) Maternal-infant outcomes: breastfeeding (initiation and continuation), infant birthweight, and post-partum pain; 3) Perinatal mental health: depression (EPDS or PHQ-9), and anxiety (GAD-7). In the sample of patients who elect to participate in IDIs, I will also assess prior trauma exposure (ACE and BTQ), PTSD symptoms (PCL-5 and City Birth Trauma Scale) and experiences of discrimination and safety in care (Personal Discrimination Multi-Item Measure).

Sample sizes for the qualitative components of the study were determined in order to achieve adequate distribution to stratify by key study variables (trauma exposure, race, pregnancy status, provider type). For the pilot implementation trial, the aim of the quantitative aims is to generate data needed to evaluate the feasibility and acceptability of the designed intervention, and to generate estimates of key parameters (variance of outcome measures) to approach power and sample size estimation for an efficacy study.

ELIGIBILITY:
Inclusion criteria for pregnant and postpartum patients for individual interviews:

* ≥ 18 years old
* under the care of an obstetrician or nurse practitioner in the U.S.,
* English-speaking
* have had ≥2 prenatal care encounters, and postpartum if they delivered a surviving infant within the past 12 months
* received care at either of the pilot sites during the pilot trial.
* Pregnant and postpartum participants will be eligible for the trauma-exposed group if they

  * report a history of trauma in childhood or adulthood,
  * are ≥1 year from the time of the traumatic experience
  * are not currently at-risk for harm from self or others
  * are willing to discuss experiences related to trauma and are able to do so without experiencing undue distress.
* Patient participants will be eligible for the non-trauma group if they deny trauma.
* Patients' stratification as White or Women of Color (any racial identity other than non-Hispanic White) will be determined by self-identification in the demographics questionnaire, rather than pre-defined groups, in order to most accurately capture participants' lived experiences.

Inclusion criteria for provider participants:

* Practicing physicians or nurses
* ≥ 6 months of experience in obstetrics
* English speaking
* Clinician Participants (providers in the participating clinics) will be enrolled in the pilot trial of the obstetric trauma-informed care toolkit intervention.
* Clinician participants will be enrolled for group or individual interviews if they consent to do so and meet above criteria.

Exclusion Criteria:

Patient participants will be excluded from the study interviews if they report

* a current unsafe environment (determined by the Assessment of Immediate Safety)
* report suicidal ideation (as determined by the PHQ9)
* report difficulty discussing experiences related to trauma.

Provider participants will be excluded from the study if they do not work at one of the pilot clinics. Provider participants will be excluded from the study interviews if they do not consent to be interviewed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Adoption of trauma-screening protocols | Change in adoption will be assessed in early implementation (2-3 months) and sustainment (6-12 months)
  The frequency with which providers assess for past and current trauma/violence will be assessed using chart review of the initial prenatal visit.
Evaluation of intervention components for adaptation and scale-up implementation | Surveys to evaluate specific components of the OB-TIC toolkit will be given in early implementation (2-3 months)
  Once the OB-TIC toolkit is complete, I will work with my mentorship team to create a survey to assess the most frequently used components of the toolkit. For example, if OB-TIC includes trauma-informed birth strategies, mental health referrals, and a modified exam procedure checklist, the survey would list each of these components and ask clinicians how often each component was used, rate how useful the component was, and whether they made changes to any of the materials.
Evaluation of intervention components for adaptation and scale-up implementation | Surveys to evaluate specific components of the OB-TIC toolkit will be given in sustainment (6-12 months)
  Once the OB-TIC toolkit is complete, I will work with my mentorship team to create a survey to assess the most frequently used components of the toolkit. For example, if OB-TIC includes trauma-informed birth strategies, mental health referrals, and a modified exam procedure checklist, the survey would list each of these components and ask clinicians how often each component was used, rate how useful the component was, and whether they made changes to any of the materials.
Change in Acceptability of Intervention Measure | Clinicians are given the survey in early implementation (2-3 months) and sustainment (6-12 months)
  Clinicians will rate acceptability on a 5-point ordinal scale ranging from "completely disagree" to "completely agree". The measure consists of 4 items and has a test-retest reliability Cronbach alpha of .83.
Change in Intervention Appropriateness Measure | Clinicians are given the survey in early implementation (2-3 months) and sustainment (6-12 months)
  Clinicians will rate appropriateness on a 5-point ordinal scale ranging from "completely disagree" to "completely agree". The measure consists of 4 items and has a test-retest reliability Cronbach alpha of .87.
Change in Feasibility of Intervention Measure | Clinicians are given the survey in early implementation (2-3 months) and sustainment (6-12 months)
  Clinicians will rate feasibility on a 5-point ordinal scale ranging from "completely disagree" to "completely agree". The measure consists of 4 items and has a test-retest reliability Cronbach alpha of .88.

SECONDARY OUTCOMES:
Change in Patient health questionnaire (PHQ-9) | The PHQ9 will be used to assess patient mood changes before (3 months prior) during (9 months) and 3 months after the pilot trial via chart review
  The PHQ-9 is a standardized measure of depression which has been used widely in obstetric settings. It consists of 9 questions and is scored from 0 to 3. Clinical significance is determined by a score of 5 or higher for mild depression and 10 or higher for moderate depression. The PHQ9 has an internal consistency of .89.
City Birth Trauma Scale | 9-12 months post-intervention
  The City Birth Trauma Scale is a 29 item scale that assesses perinatal experiences according to DSM 5 PTSD criteria. It has been shown to have reliability of .92.
Change in Appointment Adherence | Chart review will be used to assess the change in ratio of attended to scheduled appointments before (3 months prior) during (for 9 months of implementation) and after (3 months following the 9 month implementation period) the pilot trial.
  Appointment Adherence will be measured by assessing the ratio of attended to scheduled appointments. The type of appointment will also be recorded (ultrasound, initial obstetric visit, pelvic exam, medication consultation, glucose testing, etc)
Change in Elective augmentation of delivery | 3 months before the pilot, during the 9 months of implementation, and 3 months after the pilot trial assessed via chart review
  Patient preferences for augmentation of delivery will be recorded via chart review and dichotomized as yes or no.
Change Breastfeeding frequency | 3 months before the pilot, during the 9 months of implementation, and 3 months after the pilot trial assessed via chart review
  Initiation and length of continuation of breastfeeding up to 6 weeks as noted at postpartum follow-up appointment.
Change in average infant birth-weight | 3 months before the pilot, during the 9 months of implementation, and 3 months after the pilot trial assessed via chart review
  Infant birthweight as recorded in delivery note in medical record.
Change in Post-partum pain ratings | 3 months before the pilot, during the 9 months of implementation, and 3 months after the pilot trial assessed via chart review
  Postpartum pain as recorded in postpartum note in medical record.
Change in Generalized Anxiety Disorder Assessment (GAD-7) | 3 months before the pilot, during the 9 months of implementation, and 3 months after the pilot trial assessed via chart review
  The GAD-7 is a self-report measure of anxiety and worry with higher scores indicating greater severity in symptoms. The GAD-7 has demonstrated excellent internal consistency and reliability (.92).
Posttraumatic stress disorder checklist for DSM-5 (PCL-5) | After completion of the pilot trial (9-12 months after the start of implementation), a subset of patients will be recruited for interviews and completion of surveys
  The PCL-5 is a 20 item self-report measure assessing 20 post-traumatic stress disorder symptoms according to criteria in the Diagnostic and Statistical Manual (DSM-5). It has demonstrated good internal consistency and reliability (.94). A total severity score is calculated from the sum of the responses to the 20 items.
Personal Discrimination Multi- item Measure | After completion of the pilot trial, (9-12 months after the start of implementation) a subset of patients will be recruited for interviews and completion of surveys
  The PDMM a 10-item self-report measure of experiences of racism and safety in healthcare settings, with excellent reliability (.92). Responses are scored on a Likert-scale from 1 (completely disagree) to 5 (completely agree). Higher scores indicate more frequent and harmful experiences of discrimination.
Brief Trauma Questionnaire (BTQ) | After completion of the pilot trial, (9-12 months after the start of implementation) a subset of patients will be recruited for interviews and completion of surveys
  The BTQ is a 10-item self-report measure of lifetime exposure to Criterion A traumatic events. Patient participants will be asked to complete the questionnaire upon enrollment in order to determine whether they are included in the trauma group (if the score is >0) or the no-trauma group (if the score is 0).

CONTACTS AND LOCATIONS:
Overall Officials: Laura G Ward, Ph.D., Principal Investigator — The Miriam Hospital

IPD SHARING:
Plan to Share IPD: No
Since the bulk of data collected for this project are qualitative data, the decision has been made not to share these data as they may be identifying of participants.